CLINICAL TRIAL: NCT01426568
Title: A Randomised Controlled Trial of Multi-convergent Therapy for Inflammatory Bowel Disease Patients With Functional Abdominal Symptoms and High Perceived Stress
Brief Title: A Trial of Multi-convergent Therapy for Functional Symptoms and Stress in Patients With Inflammatory Bowel Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiff and Vale University Health Board (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-CMC-4876
Record Dates: First submitted 2011-08-26; First posted 2011-08-31 (Estimated); Last update posted 2020-01-30 (Actual); Status verified 2013-08

CONDITIONS: Inflammatory Bowel Disease
Keywords: Multi-Convergent Therapy; Mindfulness Meditation; Functional Abdominal Symptoms; Irritable Bowel Syndrome; Inflammatory Bowel Disease; Psychological Stress
MeSH Terms: conditions — Inflammatory Bowel Diseases; Irritable Bowel Syndrome; Stress, Psychological | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Course of Multi-Convergent Thearpy (Active Comparator)
  Interventions: Behavioral: Multi-Convergent Therapy
- Waiting List for Multi-Convergent Therapy (No Intervention)

INTERVENTIONS:
Behavioral: Multi-Convergent Therapy — Cognitive Behavioural Therapy Relaxation Techniques Meditation Stress Management
  Other Names: Mindfulness Meditation
  Arms: Course of Multi-Convergent Thearpy

SUMMARY:
The purpose of this study is to determine whether multi-convergent therapy is helpful to patients with inflammatory bowel disease who have functional abdominal symptoms or high perceived levels of psychological stress.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Inflammatory Bowel Disease
* Clinical Remission of inflammatory bowel disease as defined by an adapted disease activity index and a CRP <10
* Age 18 to 65 years
* Evidence of irritable bowel syndrome (Rome III criteria) or high perceived stress level (Levenstein perceived stress score > 0.44)

Exclusion Criteria:

* Use of steroids within 1 month of entry to study
* Initiation or change in dose of medication within 1 month of entry to the study
* Presence of ileostomy or colostomy
* Diagnosis of dementia or cognitive impairment
* Current psychosis or substance misuse
* Change in psychotropic medication in 3 months prior to entry to study
* Previous psychological interventions
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life in Inflammatory Bowel Disease Questionnaire | Assessed at baseline and at 4 months, 8 months, and 1 year

SECONDARY OUTCOMES:
Change in Irritable Bowel Syndrome Symptom Severity Score | Assessed at baseline and at 4 months, 8 months, and 1 year
Change in Levenstein Perceived Stress Score | 2 monthly intervals over 1 year
Change in Hospital Anxiety and Depression Score | 2 monthly intervals over 1 year
Abdominal Symptoms Global Improvement Score | 4 monthly intervals over 1 year
Relapse rate in inflammatory bowel disease | 1 year
Feasibility of Treatment | 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiff and Vale University Health Board, Cardiff, South Glamorgan, United Kingdom

REFERENCES:
- [Derived] Tiles-Sar N, Neuser J, de Sordi D, Baltes A, Preiss JC, Moser G, Timmer A. Psychological interventions for treatment of inflammatory bowel disease. Cochrane Database Syst Rev. 2025 Apr 17;4(4):CD006913. doi: 10.1002/14651858.CD006913.pub3. PMID 40243391
- [Derived] Berrill JW, Sadlier M, Hood K, Green JT. Mindfulness-based therapy for inflammatory bowel disease patients with functional abdominal symptoms or high perceived stress levels. J Crohns Colitis. 2014 Sep;8(9):945-55. doi: 10.1016/j.crohns.2014.01.018. Epub 2014 Feb 13. PMID 24529603